CLINICAL TRIAL: NCT01633710
Title: Protocol for a Multicentre Study to Investigate the Performance of the Padd Device in the Assessment of Peripheral Arterial Disease
Brief Title: Multicentre Study to Investigate the Performance of the Padd Device in the Assessment of Peripheral Arterial Disease
Status: Terminated | Type: Observational
Why Stopped: Redesigned sensor to be subjected to a new protocol
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Professor Kamlesh Khunti, University of Leicester
Other Study IDs: DDL-2009-01
Record Dates: First submitted 2009-07-16; First posted 2012-07-04 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-06

CONDITIONS: Peripheral Arterial Disease
Keywords: Ankle brachial pressure index; Colour duplex ultrasound; Diabetes; Photoplethysmography
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The study will compare Padd, a non-invasive automated optical device which uses a functional test to assess peripheral arterial disease (PAD), and Ankle brachial pressure index (ABPI) in the detection of PAD using as a gold standard, colour duplex ultrasound, in participants drawn from general practice, a hospital diabetic clinic and a tertiary vascular disease referral centre. The study hypothesis is that Padd performs at least as well as ABPI in detecting PAD.

DETAILED DESCRIPTION:
400 participants, with a minimum of 200 participants per site, will be recruited from two centres. At the Royal Free Hospital, London, the inclusion criterion is simply attendance at the vascular clinic; in Leicester patients >70 years or 50-69 years with a history of diabetes, smoking, known PAD or at least 2 risk factors (previous ischaemic event, hyperlipidaemia, hypertension, family history of cardiovascular disease) will be recruited from both primary care and the hospital diabetes clinic. The anticipated peripheral arterial disease detection rates are approximately 75% in London and 25% in Leicester.

In addition to standard questionnaires, participants will undergo bilateral Padd and resting ABPI. CDU will be performed by an accredited vascular technologist who will employ a scoring method consistent between both sites. The vascular technologist will be blind to the Padd and ABPI results. The results obtained with Padd and ABPI will be compared with CDU as the gold standard for this study.

The primary objectives are:

1. Performance: to compare Padd and ABPI for detecting PAD against a gold standard, CDU, performed by an experienced vascular technologist.
2. Safety: to compare adverse events using Padd, ABPI and expert CDU

The secondary objectives are:

1. to compare time taken to perform Padd and ABPI
2. to calculate specificities for Padd and ABPI
3. to investigate the impact of subject posture on the Padd results
4. to determine if skin colour has any impact on Padd performance

There are no treatments or interventions determined exclusively from the Padd readings.

ELIGIBILITY:
Inclusion criteria:

1. Royal Free Hospital - patients >50 years old referred to the vascular clinic for suspected peripheral arterial disease
2. Leicester

   * age 70 years or older
   * age 50-69 years with a history of smoking, diabetes or peripheral arterial disease
   * 50-69 years with at least two peripheral arterial disease risk factors (hyperlipidaemia, hypertension, family history of cardiovascular disease, previous ischaemic event: myocardial infarction, stroke and TIA)

Exclusion Criteria:

1. bilateral amputation that precludes placement of the Padd sensors on the feet
2. acute deep venous thrombosis, within the previous six months (application of ABPI pressure cuff on legs is not advisable for these patients)
3. skin damage or infection that precludes placement of sensors
4. active psychotic illness or severe cognitive impairment
5. inability to lie supine

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of 50 or over attending a vascular clinic at a major London hospital; patients of 70 years or over or 50-69 years with a history of diabetes, smoking, known peripheral arterial disease or at least 2 risk factors (previous ischaemic event, hyperlipidaemia, hypertension, family history of cardiovascular disease) from both primary and secondary care.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2009-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Presence or absence of peripheral arterial disease | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Kamlesh Khunti, MB BS, Principal Investigator — University of Leicester
Locations (2):
- United Kingdom (2):
  - University of Leicester, Leicester, Leicestershire
  - Royal Free Hospital, London, London